CLINICAL TRIAL: NCT03298516
Title: An Open-Label, Phase I, Dose-Escalation Study Evaluating the Safety and Tolerability of DCLL9718S in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) or DCLL9718S in Combination With Azacitidine in Patients With Previously Untreated AML Unsuitable for Intensive Induction Chemotherapy
Brief Title: A Study of DCLL9718S in Participants With Relapsed or Refractory Acute Myeloid Leukemia (AML) or DCLL9718S in Combination With Azacitidine in Participants With Previously Untreated AML Unsuitable for Intensive Induction Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO39902
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — DCLL9718S; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: DCLL9718S (Experimental): Participants will receive escalating doses of DCLL9718S intravenously (IV) in each 21-day cycle to determine MTD and RP2D in dose-escalation stage followed by DCLL9718S IV at RP2D in each 21-day cycle in dose-expansion stage until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: DCLL9718S
- Arm B: DCLL9718S and Azacitidine (Experimental): Participants will receive escalating doses of DCLL9718S (starting dose: at least one dose level below a completed and tolerated DCLL9718S monotherapy in Arm A) IV in each 28-day cycle and azacitidine 75 milligrams per square meter (mg/m^2) subcutaneously (SC) or IV on Days 1-7 of each 28-day cycle to determine MTD and RP2D of DCLL9718S in dose-escalation stage followed by DCLL9718S IV at RP2D in each 28-day cycle and azacitidine 75 mg/m^2 SC or IV on Days 1-7 of each 28-day cycle in dose-expansion stage until disease progression, unacceptable toxicity, or any other discontinuation criteria are met. Azacitidine may also be given on Days 1-5 and Days 8-9 depending on institutional preference.
  Interventions: Drug: DCLL9718S; Drug: Azacitidine

INTERVENTIONS:
Drug: DCLL9718S — DCLL9718S will be administered as per the schedule specified in the respective arm.
Drug: Azacitidine — Azacitidine will be administered as per the schedule specified in the respective arm.
  Other Names: Vidaza
  Arms: Arm B: DCLL9718S and Azacitidine

SUMMARY:
This Phase Ia/Ib, open-label, multicenter study will evaluate the safety, tolerability, and preliminary efficacy of DCLL9718S as a single agent (Phase Ia, Arm A) in participants with relapsed or refractory AML or in combination with azacitidine (Phase Ib, Arm B) in participants with previously untreated AML who are not eligible for intensive induction chemotherapy. Each arm will consist of two stages: a dose-escalation stage and an expansion stage. The dose-escalation stage is designed to establish the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D) for DCLL9718S alone (Arm A) or in combination with azacitidine (Arm B). The dose-expansion stage is designed to characterize the long-term safety and tolerability of DCLL9718S.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML per World Health Organization (WHO) criteria (except acute promyelocytic leukemia)
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Adequate end-organ function
* Willing and able to undergo a pre-treatment bone marrow aspirate and biopsy and subsequent bone marrow aspirates and biopsies during treatment

Specifically for participants in Arm A:

* Age greater than or equal to (>/=) 18 years
* Relapsed or refractory acute myeloid leukemia
* Participants cannot have received more than two prior regimens

Specifically for participants in Arm B:

* Treatment-naive participants with AML who are >/=75 years old
* Treatment-naive participants unfit for induction chemotherapy for AML due to comorbidities who are >/=65 years old

Exclusion Criteria:

* Diagnosis of acute promyelocytc leukemia
* Prior allogeneic stem cell transplant or solid organ transplant
* Active central nervous system (CNS) involvement by leukemia
* History of idiopathic pulmonary fibrosis, organizing pneumonitis (for example [e.g.], bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis
* Treatment with investigational therapy within 14 days prior to Cycle 1, Day 1
* Treatment with a monoclonal antibody within 30 days prior to Cycle 1, Day 1
* Positive for hepatitis C virus (HCV) antibody at screening
* Active hepatitis B virus (HBV) infection
* Known positivity for human immunodeficiency virus (HIV)
* History of other malignancy within 2 years prior to screening
* Family history of long QT syndrome, with a QTc interval greater than (>) 480 millisecond (msec) at screening, or taking concurrent medications known to prolong QT/QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Percentage of participants With Adverse Events (AEs) | Baseline up to end of study (up to approximately 3 years)
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Cycle 1 Day 1 up to Cycle 2 Day 1 (Cycle length: 21 days for Arm A and 28 days for Arm B)
MTD of DCLL9718S | Cycle 1 Day 1 up to Cycle 2 Day 1 (Cycle length: 21 days for Arm A and 28 days for Arm B)
RP2D of DCLL9718S | Cycle 1 Day 1 up to Cycle 2 Day 1 (Cycle length: 21 days for Arm A and 28 days for Arm B)

SECONDARY OUTCOMES:
Serum Concentration of DCLL9718S | up to 3 years
Plasma Concentration of Azacitidine | up to 3 years
Area Under the Concentration-Time Curve (AUC) of DCLL9718S | up to 3 years
Maximum Plasma Concentration Observed (Cmax) of DCLL9718S | up to 3 years
Total Clearance of DCLL9718S | up to 3 years
Terminal Half-Life (t1/2) of DCLL9718S | up to 3 years
Volume of Distribution Under Steady-State (Vss) of DCLL9718S | up to 3 years
Percentage of Participants With Complete Remission (CR), CR With Incomplete Blood Count Recovery (CRi), CR With Incomplete Platelet Count Recovery (CRp), and Overall Response, Assessed as per International Working Group (IWG) Criteria | From the date of first treatment to disease progression or relapse or death from any cause (up to approximately 3 years)
Duration of Response, Assessed as per IWG Criteria | From the date of first response to the earliest recurrence or disease progression (up to approximately 3 years)
Overall Survival | From the date of first treatment to the date of death from any cause (up to approximately 3 years)
Event-Free Survival (EFS), Assessed as per IWG Criteria | From the date of first treatment until treatment failure, relapsed from CR, CRp, or CRi, or death from any cause, whichever occurs first (up to approximately 3 years)
Progression-Free Survival (PFS), Assessed as per IWG Criteria | From the date of first treatment to disease progression or relapse or death from any cause (up to approximately 3 years)
Change From Baseline in Anti-Drug Antibody (ADA) to DCLL9718S | Baseline up to end of study (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (5):
  - City of Hope, Duarte, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Columbia University Medical Center; Research Pharmacy, Irving Pavillion, Ip 7-749, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Princess Margaret Hospital; Department of Med Oncology, Toronto, Ontario
  - Jewish General Hospital / McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Daver N, Salhotra A, Brandwein JM, Podoltsev NA, Pollyea DA, Jurcic JG, Assouline S, Yee K, Li M, Pourmohamad T, Samineni D, Sumiyoshi T, Vaze A, Dere RC, Ma C, Cooper J. A Phase I dose-escalation study of DCLL9718S, an antibody-drug conjugate targeting C-type lectin-like molecule-1 (CLL-1) in patients with acute myeloid leukemia. Am J Hematol. 2021 May 1;96(5):E175-E179. doi: 10.1002/ajh.26136. Epub 2021 Mar 11. No abstract available. PMID 33617672